CLINICAL TRIAL: NCT03596645
Title: A Phase 3 Randomized, Open-Label Study to Assess the Efficacy, Safety, and Pharmacokinetics of Golimumab Treatment, a Human Anti-TNFα Monoclonal Antibody, Administered Subcutaneously in Pediatric Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Assess the Efficacy and Safety of Golimumab in Pediatric Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: PURSUIT 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108499; CNTO148UCO3003 (Other: Janssen Research & Development, LLC); 2017-004496-31 (EudraCT Number); 2023-507142-83-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Golimumab (Experimental): Participants will receive subcutaneous (SC) golimumab through Week 50. Doses will be based on body surface area. Following the Week 54 evaluations (end of main pivotal study) participants who are benefiting from golimumab at the discretion of the investigator may continue to receive SC golimumab in an extension period until end of study.
  Interventions: Drug: Golimumab
- Group 2: Infliximab (Experimental): Participants will receive infliximab intravenous (IV) through Week 46. Doses will be based on body weight. After the Week 54 evaluations, participants receiving infliximab will be withdrawn from study participation and transition to local standard of care which may include continued commercially available infliximab at the discretion of their physician.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Golimumab — Participants receive subcutaneous (SC) golimumab through Week 50, where doses will be based on body surface area. After the Week 54 evaluations, at the discretion of investigator, participants benefiting from continued SC golimumab will continue to receive SC golimumab in the extension until end of study.
  Arms: Group 1: Golimumab
Drug: Infliximab — Participants will receive infliximab intravenous (IV) through Week 46. Doses will be based on body weight. After the Week 54 evaluations, participants receiving infliximab will be withdrawn from study participation and transition to local standard of care which may include continued commercially available infliximab at the discretion of their physician.
  Arms: Group 2: Infliximab

SUMMARY:
The purpose of this study is to evaluate efficacy of golimumab in inducing clinical remission as assessed by the Mayo score, in pediatric participants with moderately to severely active ulcerative colitis (UC). In addition, the safety profile of golimumab, in pediatric participants with moderately to severely active UC will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Must either be currently receiving treatment with, or have a history of having failed to respond to, or have a medical contraindication to at least 1 of the following therapies: oral or intravenous corticosteroids, 6-mercaptopurine, methotrexate or azathioprine OR must either have or have had a history of corticosteroid dependency (that is an inability to successfully taper corticosteroids without a return of the symptoms of ulcerative colitis [UC]) OR required more than 3 courses of corticosteroids in the past year
* Moderately to severely active UC (as defined by baseline Mayo score of 6 through 12 [endoscopy {sigmoidoscopy or colonoscopy} sub score assigned by local endoscopist], inclusive), including a (sigmoidoscopy or colonoscopy) sub score greater than or equal to (>=2)
* If receiving enteral nutrition, must have been on a stable regimen for at least 2 weeks prior to the first administration of study intervention at Week 0. Participants who receive parenteral nutrition are not permitted to enroll in the trial
* No history of latent or active tuberculosis prior to screening
* Must be up to date with all immunizations (that is, measles, mumps, rubella, and varicella) in agreement with current local immunization guidelines for immunosuppressed participants before Week 0

Exclusion Criteria:

* History of liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric (including suicidality), or metabolic disturbances
* History of malignancy or macrophage activation syndrome or hemophagocytic lymphohistiocytosis
* Have UC limited to the rectum only or to <20 percent (%) of the colon
* Presence of a stoma
* Presence or history of a fistula
* Contraindications to the use of golimumab or infliximab or anti-tumor necrosis factor (TNF-alpha) therapy per local prescribing information

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2027-02-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (58):
- United States (12):
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado and University of Colorado, Aurora, Colorado
  - Rocky Mountain Pediatric Gastroenterology, Lone Tree, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours DuPont Hospital for Children, Wilmington, Delaware
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - GI For Kids, Knoxville, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - Cook Childrens Medical Center, Fort Worth, Texas
  - DHAT Research Institute, Garland, Texas
- Belgium (3):
  - Universitair Kinderziekenhuis Koningin Fabiola, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Brussel, Jette
- Brazil (4):
  - MK Blumenau Pesquisa Clínica, Blumenau
  - Hospital Pequeno Principe, Curitiba
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - BR Trials, São Paulo
- France (2):
  - Hopital Pellegrin CHU Bordeaux, Bordeaux
  - Hôpital Necker, Paris
- Israel (6):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Assaf Harofeh Medical Center, Rishon LeZiyyon
  - Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Azienda USL di Bologna - Ospedale Maggiore, Bologna
  - AOU Meyer, Florence
  - AOU Policlinico G.Martino, Messina
  - AOU Policlinico Umberto I, Roma
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
  - Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo
  - IRCCS Materno Infantile Burlo Garofolo, Trieste
- Netherlands (2):
  - Emma Children's Hospital Academic Medical Center, Amsterdam
  - Isala Kliniek, Zwolle
- Poland (7):
  - Szpital Uniwersytecki NR 1 IM Dr Antoniego Jurasza, Bydgoszcz
  - Szpital im. M. Kopernika, Gdansk
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Wojewodzki Specjalistyczny Szpital Dzieciecy im Prof Stanislawa Popowskiego, Olsztyn
  - Korczowski Bartosz Gabinet Lekarski, Rzeszów
  - Centrum Zdrowia Matki Dziecka i Mlodziezy, Warsaw
  - Szpital Pomnik Centrum Zdrowia Dziecka, Warsaw
- South Korea (5):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp. Sant Joan de Deu, Barcelona
  - Hosp. Infantil Univ. Nino Jesus, Madrid
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Virgen Del Rocio, Seville
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital- Linkou, Taoyuan

REFERENCES:
- [Derived] Turner D, Lomax KG, Veereman G, Griffiths AM, Kierkus J, Kang B, Berezny K, Padgett L, Mao G, Zitser Y, Strauss RS, Verhoeven J, Adedokun OJ, Hyams JS. Efficacy, Safety, and Pharmacokinetics of Golimumab in Children with Moderately-To-Severely Active Ulcerative Colitis: Results from the PURSUIT 2 Study. Inflamm Bowel Dis. 2026 Jan 8:izaf322. doi: 10.1093/ibd/izaf322. Online ahead of print. PMID 41503939

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results are currently reported until the primary completion date (21-Nov-2023). Final results will be posted upon study completion.
Groups:
- Group 1: Golimumab: In short term phase (Week 0-6), participants weighing greater than or equal to (>=) 45 kilograms (kg), received fixed subcutaneous induction doses of golimumab 200 milligrams (mg) at Week 0 and 100 mg at Week 2. Participants weighing less than (<) 45 kg received body surface area (BSA) adjusted doses with 120 milligrams per square meter (mg/m^2) (up to a maximum of 200 mg) at Week 0 and 60 mg/m^2 (up to a maximum of 100 mg) at Week 2. In long-term Phase (Week 6 through Week 54), participants who showed a clinical response at Week 6 continued receiving subcutaneous golimumab 100 mg or 60 mg/m^2 every 4 weeks (q4w) through Week 50. Participants with no clinical response (non-responders) at Week 6 received additional golimumab doses at Weeks 6 and 10 at the discretion of the investigator. Participants who showed partial Mayo response at Week 14, continued golimumab 100 mg or 60 mg/m^2 qw4 through Week 50. Participants without a partial Mayo response at Week 14 were withdrawn from further treatment and entered a 16-week safety follow-up period after the last dose. In study extension (Week 54 to end of study) phase, participants who were benefited from golimumab, at the discretion of the investigator, continued to receive SC golimumab q4w until marketing authorization is obtained for golimumab or participant turns 18 years had access to commercially available golimumab or decided by the sponsor.
- Group 2: Infliximab: In short term phase (Week 0-6), participants weighing >=30 kg, received infliximab 5 mg/kg intravenous (IV) infusion at Week 0 and Week 2. In long-term Phase (Week 6 through Week 54), participants who showed a clinical response at Week 6 continued to receive infliximab 5 mg/kg IV infusion every 8 weeks (q8w) through Week 46. Participants who did not show a clinical response at Week 6 received an increased dose of infliximab that is 10 mg/kg (capped at 1 gram) starting at Week 6 and every q8q thereafter, or 5 mg/kg at Week 6 and Week 8 followed by 10 mg/kg (capped at 1 gram) at Week 14 and every q8w thereafter. Participants who showed a partial Mayo responders at Week 14 continued infliximab 10 mg/kg every 8 weeks through Week 46. Participants who did not show partial Mayo response at Week 14 either received a further dose escalation to 10 mg/kg q4w (capped at 1 gram) or were withdrawn from the study. At Week 22, participants who received the escalated dose of infliximab 10 mg/kg q4w were required to show a partial Mayo response and who met this criterion continued to receive open-label infliximab 10 mg/kg (capped at 1 gram) q4w through Week 50. After Week 54 evaluations, participants receiving infliximab were withdrawn from study participation and transitioned to local standard of care.
Period: Overall Study
Arm/Group | Group 1: Golimumab | Group 2: Infliximab
Started | 69 | 15
Treated | 69 | 14
Completed | 0 | 0
Not Completed | 69 | 15
Not completed — Adverse Event | 17 | 0
Not completed — Lack of Efficacy | 8 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Initiated Prohibited Medication | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 0
Not completed — No mucosal healing achieved | 1 | 0
Not completed — Disease progression | 1 | 0
Not completed — Ongoing | 37 | 12
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Group 1 Golimumab arm: Full Golimumab analysis set 1 (FGAS1) included all enrolled participants who received at least 1 dose (complete or partial) of golimumab during the Short-Term Phase (Weeks 0-6). Group 2: Infliximab arm: Full Infliximab analysis set 1 (FIAS1) included all enrolled participants who received at least 1 dose (complete or partial) of infliximab during the Short-Term Phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Golimumab | Group 2: Infliximab | Total
Number analyzed (Participants) | 69 | 14 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.4 (3.3) | 14.3 (2.23) | 13.6 (3.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 8 | 45
  Male | 32 | 6 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 0 | 17
  Not Hispanic or Latino | 50 | 14 | 64
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 12 | 5 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 50 | 9 | 59
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 3 | 0 | 3
  Brazil | 11 | 0 | 11
  France | 1 | 0 | 1
  Israel | 10 | 3 | 13
  Italy | 9 | 2 | 11
  Poland | 16 | 3 | 19
  Korea, South | 12 | 5 | 17
  Spain | 3 | 0 | 3
  United States | 4 | 1 | 5
Age Categorical [Count of Participants; unit: Participants]
  2-5 years | 2 | 0 | 2
  6-11 years | 13 | 2 | 15
  12-17 years | 54 | 12 | 66

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Remission at Week 6 as Assessed by the Mayo Score
Description: Percentage of participants with clinical remission at Week 6 as assessed by the Mayo score was reported. Clinical remission was defined as a Mayo score of less than or equal to (<=) 2 point, with no individual sub-score greater than (>) 1. The Mayo score was sum of 4 sub-scores (that is, stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total score was calculated as the sum of the 4 sub scores and values ranged from 0 to 12. A score of 3 to 5 points indicated mildly active disease; a score of 6 to 10 indicated moderately active disease; and a score of 11 to 12 indicated severe disease.
Time Frame: Week 6
Population: FGAS1 included all enrolled participants who received at least 1 dose (complete or partial) of golimumab during the induction phase. This outcome measure was planned to be reported for "Group 1: Golimumab" arm only.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Golimumab
Number analyzed (Participants) | 69
Percentage of participants | 31.9 [22.7 to 41.1]

2. Secondary Outcome: Percentage of Participants With Symptomatic Remission at Week 54
Description: Percentage of participants with symptomatic remission at Week 54 was reported. Symptomatic remission was defined as a Mayo stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0. Mayo stool frequency subscore was determined on the average number of stools more than normal in 24 hours, score ranged from 0 (normal number of stools) to 3 (5 or more stools more than normal), higher score indicated more severity. Mayo rectal bleeding subscore ranged from 0 (no blood seen) to 3 (blood alone passed), higher score indicated more severity.
Time Frame: Week 54
Population: Full golimumab analysis set 2 (FGAS2) included participants who were in clinical response at Week 6 to golimumab as assessed by the Mayo score (local reader) and who received at least 1 dose (complete or partial) of golimumab during the long-term phase. This outcome measure was planned to be reported for "Group 1: Golimumab" arm only.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Golimumab
Number analyzed (Participants) | 41
Percentage of participants | 39.0 [26.5 to 51.6]

3. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 54 as Assessed by the Mayo Score
Description: Percentage of participants with clinical remission at Week 54 was reported. Clinical remission was defined as a Mayo score <= 2 points, with no individual subscore >1. The Mayo score was the sum of 4 sub-scores (that is, stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total score was calculated as the sum of the 4 sub scores and values ranged from 0 to 12. A score of 3 to 5 points indicated mildly active disease; a score of 6 to 10 indicated moderately active disease; and a score of 11 to 12 indicated severe disease.
Time Frame: Week 54
Population: FGAS2 included participants who were in clinical response at Week 6 to golimumab as assessed by the Mayo score (local reader) and who received at least 1 dose (complete or partial) of golimumab during the long-term phase. This outcome measure was planned to be reported for "Group 1: Golimumab" arm only.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Golimumab
Number analyzed (Participants) | 41
Percentage of participants | 31.7 [19.8 to 43.7]

4. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 54 as Assessed by the Pediatric Ulcerative Colitis Activity Index Score (PUCAI) Score
Description: Percentage of participants with clinical remission at Week 54 as assessed by PUCAI score was reported. Clinical remission as measured by the PUCAI score was a PUCAI score <10. PUCAI score was intended for pediatric participants with UC. PUCAI consisted of the following 6 subscores with scores as: abdominal pain (no pain =0, pain can be ignored =5, pain cannot be ignored =10); rectal bleeding (none =0, small amount only [in less than 50 percent (%) of stools] =10, small amount with most stools =20, large amount [>50% of the stool content] =30); stool consistency of most stools (formed =0, partially formed =5, completely unformed =10); number of stools per 24 hours (0-2 =0, 3-5 =5, 6-8 =10, >8 =15); nocturnal bowel movement (no =0, yes =10); activity level (no limitation of activity =0, occasional limitation of activity =5, severely restricted activity =10). PUCAI score = sum of scores of 6 items; score range of 0= no severity to 85= extreme severity.
Time Frame: Week 54
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Golimumab
Number analyzed (Participants) | 41
Percentage of participants | 34.1 [22.0 to 46.3]

5. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 6 as Assessed by the Pediatric Ulcerative Colitis Activity Index Score (PUCAI) Score
Description: Percentage of participants with clinical remission at Week 6 as assessed by PUCAI score was reported. Clinical remission as measured by the PUCAI score was a PUCAI score <10. PUCAI score was intended for pediatric participants with UC. PUCAI consisted of the following 6 subscores with scores as: abdominal pain (no pain =0, pain can be ignored =5, pain cannot be ignored =10); rectal bleeding (none =0, small amount only [in less than 50% of stools] =10, small amount with most stools =20, large amount [>50% of the stool content] =30); stool consistency of most stools (formed =0, partially formed =5, completely unformed =10); number of stools per 24 hours (0-2 =0, 3-5 =5, 6-8 =10, >8 =15); nocturnal bowel movement (no =0, yes =10); activity level (no limitation of activity =0, occasional limitation of activity =5, severely restricted activity =10). PUCAI score = sum of scores of 6 items; score range of 0= no severity to 85= extreme severity.
Time Frame: Week 6
Population: FGAS1 included all enrolled participants who received at least 1 dose (complete or partial) of golimumab during the Short-Term Phase (Weeks 0-6). This outcome measure was planned to be reported for "Group 1: Golimumab" arm only.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Golimumab
Number analyzed (Participants) | 69
Percentage of participants | 33.3 [24.0 to 42.7]

6. Secondary Outcome: Percentage of Participants With Clinical Response at Week 6 as Assessed by the Mayo Score
Description: Clinical response was defined as a decrease from baseline in the Mayo score by >= 30% and >= 3 points, with either a decrease from baseline in the rectal bleeding subscore of >= 1 or a rectal bleeding subscore of 0 or 1. The Mayo score was the sum of 4 sub-scores (that is, stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total score was calculated as the sum of the 4 sub scores and values ranged from 0 to 12. A score of 3 to 5 points indicated mildly active disease; a score of 6 to 10 indicated moderately active disease; and a score of 11 to 12 indicated severe disease.
Time Frame: Week 6
Population: as for outcome 5
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Golimumab
Number analyzed (Participants) | 69
Percentage of participants | 56.5 [46.7 to 66.3]

7. Secondary Outcome: Percentage of Participants With Endoscopic Healing at Week 6 as Assessed by the Mayo Score
Description: Percentage of participants with endoscopic healing at Week 6 as assessed by the Mayo score was reported. Endoscopic healing was defined by an endoscopy subscore of the Mayo score of 0 or 1 based on local endoscopy. The Mayo score was the sum of 4 sub-scores (that is, stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each subscore rated on a scale from 0 (normal) to 3 (severe), with higher scores indicating more severe disease. The total score was calculated as the sum of the 4 sub scores and values ranged from 0 to 12. A score of 3 to 5 points indicated mildly active disease; a score of 6 to 10 indicated moderately active disease; and a score of 11 to 12 indicated severe disease.
Time Frame: Week 6
Population: as for outcome 5
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Golimumab
Number analyzed (Participants) | 69
Percentage of participants | 40.6 [30.9 to 50.3]

8. Secondary Outcome: Percentage of Participants With Endoscopic Healing at Week 54 as Assessed by the Mayo Score
Description: Percentage of participants with endoscopic healing at Week 54 as assessed by the Mayo score was reported. Endoscopic healing is defined as an endoscopy subscore of the Mayo score of 0 or 1 based on local endoscopy. The Mayo score was the sum of 4 sub-scores (that is, stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each subscore rated on a scale from 0 (normal) to 3 (severe), with higher scores indicating more severe disease. The total score was calculated as the sum of the 4 sub scores and values ranged from 0 to 12. A score of 3 to 5 points indicated mildly active disease; a score of 6 to 10 indicated moderately active disease; and a score of 11 to 12 indicated severe disease.
Time Frame: Week 54
Population: FGAS2 included participants who were in clinical response at Week 6 to golimumab as assessed by the Mayo score (local reader) and who received at least 1 dose (complete or partial) of golimumab during the long-term phase. This outcome measure was planned to be analyzed for "Group 1: Golimumab" arm only.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Golimumab
Number analyzed (Participants) | 41
Percentage of participants | 36.6 [24.2 to 49.0]

9. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 54 as Assessed by the Mayo Score for Participants Who Were in Clinical Remission at Week 6
Description: Percentage of participants with clinical remission at Week 54 as assessed by the Mayo score for participants who were in clinical remission at week 6 was reported. Clinical remission was defined as a Mayo score <=2 points, with no individual subscore >1. The Mayo score was the sum of 4 sub-scores (that is, stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total score was calculated as the sum of the 4 sub scores and values ranged from 0 to 12. A score of 3 to 5 points indicated mildly active disease; a score of 6 to 10 indicated moderately active disease; and a score of 11 to 12 indicated severe disease.
Time Frame: Week 54
Population: Analysis population included participants who had achieved clinical remission at Week 6. This outcome measure was planned to be reported for "Group 1: Golimumab" arm only.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Golimumab
Number analyzed (Participants) | 22
Percentage of participants | 54.5 [37.1 to 72.0]

10. Secondary Outcome: Percentage of Participants Who Were Not Receiving Corticosteroids for at Least 12 Weeks Prior to Week 54 and in Clinical Remission at Week 54
Description: Percentage of participants who were not receiving corticosteroids for at least 12 weeks prior to Week 54 and in clinical remission at week 54 was reported. Clinical remission was defined as a Mayo score <=2 points, with no individual subscore >1. The Mayo score was the sum of 4 sub-scores (that is, stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment); each rated on a scale from 0 to 3, with higher scores indicating more severe disease. The total score was calculated as the sum of the 4 sub scores and values ranged from 0 to 12. A score of 3 to 5 points indicated mildly active disease; a score of 6 to 10 indicated moderately active disease; and a score of 11 to 12 indicated severe disease.
Time Frame: Week 54
Population: as for outcome 8
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Golimumab
Number analyzed (Participants) | 41
Percentage of participants | 31.7 [19.8 to 43.7]

ADVERSE EVENTS:
Time Frame: All cause mortality: From screening (-6 weeks) up to Week 70; serious adverse events (SAEs) and other adverse events (AEs): From baseline (Day 1) up to Week 70
Description: (Group 1: Golimumab) arm: Safety Golimumab analysis set included all enrolled participants who received at least 1 dose (complete or partial) of golimumab. (Group 2: Infliximab arm): Safety Infliximab analysis set includes all enrolled participants who received at least 1 dose (complete or partial) of infliximab.
Arm/Group | Group 1: Golimumab | Group 2: Infliximab
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/14
Serious Adverse Events (participants affected / at risk) | 28/69 | 2/14
Other Adverse Events (participants affected / at risk) | 62/69 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Golimumab (N=69) | Group 2: Infliximab (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 17 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 1 | 0
Covid-19 (Infections and infestations) | 1 | 0
Cytomegalovirus Colitis (Infections and infestations) | 2 | 0
Cytomegalovirus Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Pseudomembranous Colitis (Infections and infestations) | 1 | 0
Stump Appendicitis (Infections and infestations) | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fungal Test Positive (Investigations) | 1 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast Mass (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Golimumab (N=69) | Group 2: Infliximab (N=14)
Anaemia (Blood and lymphatic system disorders) | 10 | 3
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 8 | 5
Colitis Ulcerative (Gastrointestinal disorders) | 31 | 7
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 7 | 1
Mucous Stools (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1
Fatigue (General disorders) | 4 | 0
Pyrexia (General disorders) | 7 | 3
Covid-19 (Infections and infestations) | 13 | 1
Cystitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 5 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1
Pharyngitis (Infections and infestations) | 3 | 1
Respiratory Tract Infection (Infections and infestations) | 5 | 0
Rhinitis (Infections and infestations) | 3 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 13 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1
Faecal Calprotectin Increased (Investigations) | 3 | 0
Weight Decreased (Investigations) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 12 | 2
Renal Cyst (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Acne (Skin and subcutaneous tissue disorders) | 7 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-11-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03596645/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT03596645/SAP_001.pdf